CLINICAL TRIAL: NCT00436657
Title: A Phase I Study of Continuous Hyperthermic Peritoneal Perfusion (CHPP) With Escalating Doses of Cisplatin for Children With Peritoneal Carcinomatosis or Advanced Peritoneal and Retroperitoneal Disease
Brief Title: Continuous Hyperthermic Peritoneal Perfusion (CHPP) With Cisplatin for Children With Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0917
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Peritoneal Neoplasms; Retroperitoneal Neoplasms; Gastrointestinal Neoplasms; Adenocarcinoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Adrenocortical Carcinoma; Wilms Tumor; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor
Keywords: Children; Pediatric; Peritoneal Tumor; Retroperitoneal Tumor; Gastrointestinal Adenocarcinoma; Desmoplastic Round Cell Tumor; Neuroblastoma; Ovarian Germ Cell; Sarcoma; Adrenocorticocarcinoma; Wilms' Tumor; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor; Recurrent Tumors; Cisplatin; Platinol®-AQ; Platinol®; CDDP; Abdominal Wash; Hyperthermic Perfusion; Continuous Hyperthermic Peritoneal Perfusion; CHPP
MeSH Terms: conditions — Peritoneal Neoplasms; Retroperitoneal Neoplasms; Gastrointestinal Neoplasms; Adenocarcinoma; Neuroblastoma; Ovarian Neoplasms; Sarcoma; Adrenocortical Carcinoma; Wilms Tumor; Rhabdomyosarcoma; Desmoplastic Small Round Cell Tumor; Neoplasms | interventions — Cisplatin; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery + CHPP of Escalating Cisplatin (Experimental): Abdominal Surgery + CHPP of Escalating Cisplatin (Starting dose of 100 mg/m^2 intraperitoneally delivered as Continuous Hyperthermic Peritoneal Perfusion (CHPP) over 90 minutes at a flow rate of 1.5L/min and a peritoneal temperature of 42.5°Celsius.)
  Interventions: Drug: CHPP of Cisplatin; Procedure: Abdominal Surgery

INTERVENTIONS:
Drug: CHPP of Cisplatin — Starting dose of 100 mg/m^2 intraperitoneally delivered as Continuous Hyperthermic Peritoneal Perfusion (CHPP) over 90 minutes at a flow rate of 1.5L/min and a peritoneal temperature of 42.5°Celsius.
  Other Names: Platinol®-AQ; Platinol®; CDDP; Abdominal Wash; hyperthermic perfusion
Procedure: Abdominal Surgery — Surgical removal of abdominal tumors.
  Other Names: cytoreductive surgery

SUMMARY:
There has been no successful treatment of diffuse peritoneal metastasis or carcinomatosis, in childhood tumors. Once this advanced stage of disease is evident, survival is measured in weeks. The selective lethal effect of supranormal temperatures on neoplastic cells and the additive or synergistic effect of combining chemotherapy has been well established in adult clinical trials using continuous hyperthermic peritoneal perfusion (CHPP) for advanced peritoneal adenocarcinoma of gastrointestinal origin, ovarian carcinoma and mesothelioma.

This phase I study will evaluate the safety of continuous hyperthermic peritoneal perfusion with escalating doses of intraperitoneal cisplatin in the treatment of children with refractory tumors limited to the abdominal cavity. If tumors are outside the abdominal cavity, the tumors must be able to be controlled.

Since CHPP has potential to improve outcome of children with peritoneal and retroperitoneal metastases, this study will evaluate the safety of elevated temperature (40oC) with intraperitoneal cisplatin chemotherapy.

Primary Objectives:

1. To determine the MTD and dose-limiting toxicity of intraperitoneal cisplatin given in combination with CHPP as a 90 minute perfusion in children with advanced peritoneal and retroperitoneal solid tumors
2. To determine the safe and tolerable dose of CHPP with cisplatin to be used in Phase II trials
3. To determine the pharmacokinetics of intraperitoneal cisplatin platinum given with CHPP as a 90 minute abdominal perfusion (Optional)

DETAILED DESCRIPTION:
Cisplatin has an atom at its center that contains platinum. The platinum is supposed to poison the cancer cells, causing them to eventually die. Sodium thiosulfate is designed to bind-up any Cisplatin that has escaped from the abdomen into the blood stream.

This is an investigational treatment which has been performed on two children on a compassionate use basis in North America. Both surgeries were performed at M.D. Anderson by the Study Chairman.

Before you can start receiving the study drugs, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. A physical exam will be performed, and you will have a computed tomography (CT) scan, or magnetic resonance imaging (MRI) scan to make sure the disease is only in the abdomen (stomach area). Blood (about 1 teaspoon) will be drawn for routine tests. You may have an echocardiogram (ECHO--a test to check heart function), and electrocardiogram (ECG--a test to measure electrical activity of the heart) if you have ever taken an anthracycline drug. An echocardiogram uses sound waves to make pictures of your heart, which helps show how well your heart pumps blood. You will be asked to lie on your left side while a technician places a probe with gel on your chest to create images of your heart to determine the function and size. Women who are able to have children must have a negative urine pregnancy test.

If you are found to be eligible, you will have a hearing test before your surgery and at your one-month evaluation.

If you are found to be eligible, the abdominal surgery will be performed to try to remove as many tumors as possible. The surgeon may decide during the surgery that the abdominal wash will not be performed, for example if the disease has spread to or attached to certain organs. If this occurs, your doctor will discuss other treatment options with you.

If the doctor decides that you are eligible to receive the abdominal wash, a drug called sodium thiosulfate will be given through a needle in your vein. The abdomen will then be temporarily closed. Then the abdominal wash will begin. This will be done in the same room while you are under anesthesia. During the "abdominal wash," the heated cisplatin will be given into your abdomen and will "wash" over the area of the surgical procedure. There will be a pump attached to the plastic tubing and that will pump the drug in and out of your abdomen during that 90 minute period while the surgeon is gently compressing your abdominal wall so that the drug can reach all areas of your abdomen equally. After 90 minutes the drug is removed and your abdomen is 'washed' with saline. Then all the fluid is removed and the surgeon permanently closes your abdomen with 3 layers of stitches.

The actual dose level of cisplatin that you will receive will be decided when you enter the study. Participants on this study will be enrolled in groups of 3, and each group will be given a specific dose level of cisplatin. The first group will receive the lowest dose of cisplatin. If there are no severe or life-threatening side effects in this first group of patients, the next group will receive a higher dose of cisplatin and so on. This process of increasing the dose level for each new group of participants will continue until some patients have severe or life-threatening side effects. At that point, the dose level of cisplatin will be lowered and tested again in more participants.

Blood (about 1 teaspoon) will be drawn for routine tests. This testing will take place during the operation and every day until you leave the hospital.

After you leave the hospital, you will have a study visit about 1 month later, and then every 3 months for 6 months. At these visits, you will have a CT scan or MRI scan and a physical exam to check the status of the disease.

You will be taken off study if the disease gets worse or if you are disease free at or after your 6 month follow-up.

This is an investigational study. Cisplatin is FDA-approved and commercially available. Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 3 and less than or equal to 18 years
2. Histologically proven diffuse peritoneal or retroperitoneal tumor from the following histologies: adenocarcinoma of the gastrointestinal tract, desmoplastic round cell tumor, late stage neuroblastoma, ovarian germ cell, sarcoma, adrenocorticocarcinoma, Wilms', rhabdomyosarcoma. (target groups: desmoplastic small round cell tumor (DSRCT), neuroblastoma, and recurrent tumors). If tumors are outside the abdominal cavity, the tumors must be controllable.
3. All patients must have refractory or recurrent tumors with no known curative treatment options.
4. Radiologic workup must demonstrate that the disease is confined to the abdominal cavity. If tumors are outside the abdominal cavity, the tumors must be able to be controlled.
5. Radiologic workup or prior abdominal exploration must be consistent with disease which can be debulked to a residual size of less than or equal to 1 mm thickness per tumor deposit
6. Patients must have minimum expected duration of survival of greater than 6 weeks
7. Patients must not have any systemic illness which precludes them from being an operative candidate. This includes but is not limited to sepsis, liver failure, pregnancy, lactating females.
8. Patients must have fully intact mental status and normal neurologic abilities.
9. Patients must have adequate renal function (serum creatinine </= 1.5 without history dialysis or renal failure)
10. Patients will be eligible if the white blood count (WBC) is > or =2,000/ul or Absolute neutrophil count (ANC) is > or =1,500, or platelets are > or = 100,000/mm^3
11. Patients will be eligible if serum total bilirubin and liver enzymes (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) are </= 2 times the upper limit of normal
12. Patients must be recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy and be at least 14 days past the date of their last treatment
13. If tumors are outside the abdominal cavity, the tumors must be controllable.

Exclusion Criteria:

1. Patients who have failed previous continuous hyperthermic intraperitoneal perfusion with platinum therapy will be ineligible
2. Patients with tumors that are unable to be controlled outside the abdominal cavity will be ineligible
3. Patients will be ineligible if they have any concomitant cardiopulmonary disease which would place them at unacceptable risk for a major surgical procedure
4. Patients will be ineligible if they have a baseline neurologic toxicity of Grade 3 or greater (because of the potential neurotoxicity associated with platinum)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of continuous hyperthermic peritoneal perfusion (CHPP) with cisplatin in children with peritoneal cancer | Assessed during treatment and post surgery through hospital stay (estimated 5 days) followed one month later.
  The MTD is defined as the highest dose in which 1 or fewer patients in 6 treated experience a dose limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hayes-Jordan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org